CLINICAL TRIAL: NCT01984489
Title: A Multicenter Randomized, Double-blind, Placebo Controlled ,Parallel Group ,Phase II Study to Access the Efficacy and Safety of SHR117887 in Combination Therapy With Metformin in Patients With Type 2 Diabetes Patients
Brief Title: Efficacy and Safety Study of SHR117887 in Combination With Metformin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR117887-201
Record Dates: First submitted 2013-11-08; First posted 2013-11-14 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Type 2 Diabetes
Keywords: SHR117887, Metformin,combination,PhaseII
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo/Metformin (Placebo Comparator): patients are administered oral tablets of placebo once daily and 500mg TID for 4 weeks at the run-in period. After randomized ,patients administer the drugs too.
  Interventions: Drug: Placebo
- SHR117887 (50mg q.d)/Metformin (Experimental): patients are administered oral placebo once daily and metformin 500mg TID for 4 weeks at the run-in period.After randomised,patients adminitered SHR117887 50mg QD and metformin 500mg TID for 12 weeks.
  Interventions: Drug: SHR117887
- SHR117887 (100mg q.d)/Metformin (Experimental): patients are administered oral placebo once daily and metformin 500mg TID for 4 weeks at the run-in period.After randomised,patients adminitered SHR117887 100mg QD and metformin 500mg TID for 12 weeks.
  Interventions: Drug: SHR117887

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo/Metformin
Drug: SHR117887
  Arms: SHR117887 (100mg q.d)/Metformin; SHR117887 (50mg q.d)/Metformin

SUMMARY:
SHR117887 is a new dipeptidyl peptidase(DPP)-4 inhibitor. This study aims to evaluate the efficacy and safety of SHR117887 in combination therapy with Metformin in patients with Type 2 Diabetes in Metformin monotherapy Who have Inadequate Glycemic Control

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 2 diabetes mellitus
* Patients have been treated with metformin for at least 8 weeks and be on a stable dose of at least 1500mg daily prior to the screening visit
* HbA1C：≥7.5% and ≤11.0% at screeing visit and at the end of run-in period
* Age:≥20 and ≤70 years
* BMI(body mass index):≥20 and ≤35 kg/m2

Exclusion Criteria:

-

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in HbA1c (Hemoglobin A1C) at Week 12 | 12 weeks

SECONDARY OUTCOMES:
Percentage of Participants Achieving Less Than (<) 6.5% or <7% HbA1c Levels | 12 weeks
Change From Baseline in Fasting Plasma Glucose,insulin and C-peptide at Week 12 | 12 weeks
Post-meal total and incremental glucose,insulin and C-peptide area under the curve at week 12 | 12 weeks
Change From Baseline in Body Weight at Week 12 | 12 weeks